CLINICAL TRIAL: NCT01407549
Title: The Influence of Mindfulness Based Intervention on Pain Perception in Chronic Pain Patients Evaluating Personal Characteristics and Possible Mechanism
Brief Title: The Influence of Mindfulness Based Intervention on Pain Perception in Chronic Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMC11114119KCTIL
Record Dates: First submitted 2011-07-26; First posted 2011-08-02 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2012-06

CONDITIONS: Low Back Pain; Osteoarthritis
MeSH Terms: conditions — Low Back Pain; Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): The intervention group will participate in the Mindfulness Program consists of one 2-hour session each week for 6 consecutive weeks plus a half day retreat near the end of the intervention.
  Interventions: Behavioral: mindfulness group meetings with psychologist
- Control group (No Intervention): Participants in the control group will be assigned to a waiting list group. Participants will be told that they will be eligible for the intervention three months after the completion of a preliminary documentation of their symptoms and additional measures. Participants will complete the same battery of measures according to the same time table as participants in the intervention group.

INTERVENTIONS:
Behavioral: mindfulness group meetings with psychologist — The Mindfulness Program consists of one 2-hour session each week for 6 consecutive weeks plus a half day retreat near the end of the intervention. Participants will attend weekly group meetings (15-20 individuals per group) in which they will be guided through a progressive experiential exploration of mindfulness. Participants will be asked to develop a daily meditation practice of 30-45 minutes with audio-recordings for guidance, and will report the amount and type of practice in a daily dairy. . A psychologist with rich personal experience in mindfulness who is trained in mindfulness based therapy will be responsible for administering the program.
  Arms: Intervention group

SUMMARY:
Background: Chronic pain is a common condition in the general population, causing great suffering in both physical and mental aspects. Previous research shows that mindfulness based interventions help chronic pain patients to cope better with their pain, and improve their quality of life. Although evidence support the efficacy of mindfulness based interventions for chronic pain, it is still unclear whether this efficacy involves a direct influence on sensory aspects of pain perception. Further more, the mechanisms of change responsible for the improved life quality and the possible moderating factors that may influence treatment efficacy, are still unknown.

Aim: The purpose of this study is to evaluate the efficacy of mindfulness based intervention on pain perception and quality of life in individuals suffering from chronic pain. The investigators will also evaluate potential mechanisms responsible for the change following mindfulness practice. Finally the investigators will examine the role of personal characteristics as potential moderating factors of mindfulness effect.

Hypothesis: The investigators hypothesize that 1) compared to a waitlist control group, chronic pain patients participating in a full mindfulness based program will report greater improvements in a) pain severity, b) quality of life and psychological symptoms, and c) will demonstrate changes in physiological characteristics of pain. 2) Changes following the mindfulness based program will be mediated by change in pain catastrophizing, self regulation capacity and pain acceptance. 3) The investigators hypothesize that gender, baseline mindfulness, and anxiety sensitivity will moderate the efficacy of the mindfulness based program.

Method: A randomized controlled design will be used to evaluate the efficacy of mindfulness based intervention on pain perception and quality of life in individuals suffering from chronic recurrent low back pain and osteoarthritis. Participants will be randomized to a mindfulness based treatment group, or to a waitlist control group, and will be assessed for psychological variables and psychophysical pain assessment before treatment. Participants allocated to treatment group will then attend six group meetings in which they will learn and practice different mindfulness meditation techniques, and will be asked to practice these techniques on a daily basis. Post treatment assessments will take place at the end of the intervention for both treatment and control groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who suffer from recurrent chronic low back pain
2. Patients who suffer from osteoarthritis pains.
3. The pain has to be persistent for 3 months or longer and at least moderate in severity.

Exclusion Criteria:

1. mental illness with psychotic features
2. cognitive impairment
3. a history of an inpatient admission for psychiatric disorder within the past two years
4. diagnosis of a life threatening medical condition (e.g., cancer)
5. patients who are planning to start using other types of alternative interventions parallel to the Mindfulness Program.

Ages: 24 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
change in Brief Pain Inventory Short Form questionnaire (BPI-sf) | Administration will take place upon entry into the study, after 4 weeks of participating in the program, and at the completion of the 6-weeks programs. Follow up of psychological measures will be held 3 months after completing the program by telephone.
  measures and characterize pain and the interference of pain with the patient's life (reactive dimension). The BPI questionnaire includes a 0-10 rating scale to measure the pain and the influence of pain on different aspects of daily life (general activity, mood, sleep, relationship with other people, work) that constitute the life impact index

SECONDARY OUTCOMES:
Brief Symptom Inventory (BSI) | upon entry into the study, after 4 weeks of participating in the program, and at the completion of the 6-weeks programs. Follow up of psychological measures will be held 3 months after completing the program by telephone.
  53 items and provides nine sub-scale scores measuring a range of psychological symptoms and somatic complaints. Participants rate on a scale of 0 ('not at all') to 4 ('extremely') how much they were bothered in the last 7 days by each of 18 symptoms, including separate scores for anxiety, depression, somatization, and a global symptom severity index
SF-12 Quality of life | upon entry into the study, after 4 weeks of participating in the program, and at the completion of the 6-weeks programs. Follow up of psychological measures will be held 3 months after completing the program by telephone.
  The Short-Form General Health Survey is a shorter form of the widely used SF-36 and assesses health-related quality of life. It consists of 12 items that allow the calculation of 'physical health' (PCS-12) and 'mental health' (MCS-12) summary scales.
Psychophysical measures | at the entry into the study, and after 6 weeks
  Using the The Thermal Sensory Analyzer we will measure Heat/ Cold pain threshold (HPT/CPT)and Supra threshold pain.
The Pain Catastrophizing Scale | upon entry into the study, after 4 weeks of participating in the program, and at the completion of the 6-weeks programs. Follow up of psychological measures will be held 3 months after completing the program by telephone.
  Sullivan, Bishop, & Pivik, 1995) This questionnaire includes 13 items representing the three components of pain catastrophizing: rumination (e.g., "I can't seem to keep it out of my mind"); magnification (e.g., "I wonder whether something serious may happen"); and helplessness (e.g., "There is nothing I can do to reduce the intensity of pain").
Difficulties in Emotion Regulation Scale (DERS) | upon entry into the study, after 4 weeks of participating in the program, and at the completion of the 6-weeks programs. Follow up of psychological measures will be held 3 months after completing the program by telephone.
  consists of 36 self-report items which comprise six subscales that investigate individuals' complaints about emotional regulation problems. The scales are: Non-acceptance of Emotional Response, Difficulties engaging in Goal-Directed Behavior, Impulse Control Difficulties, Lack of Emotional Awareness, limited access to Emotion Regulation Strategies and Lack of Emotional Clarity. Respondents are asked to rate their self-perceptions regarding each item on a 5-point Likert scale, which ranges from "almost never" to "almost always."
The Chronic Pain Acceptance Questionnaire (CPAQ) | upon entry into the study, after 4 weeks of participating in the program, and at the completion of the 6-weeks programs. Follow up of psychological measures will be held 3 months after completing the program by telephone.
  a 20-item, two factor (Activity Engagement and Pain Willingness) questionnaire, adapted through the process of factor analysis from the original, longer version (Geiser, 1992).
Anxiety Sensitivity Index (ASI) | at the entry into the study, and after 6 weeks
  a 16-item measure on which respondents indicate, on a 5-point Likert-type scale (0=very little to 4=very much), the degree to which they fear the potential negative consequences of anxiety-related symptoms and sensations. The ASI is made up of one higher-order factor (ASI total score) and three lower-order factors: Physical, Psychological, and Social Concerns
Mindful Attention Awareness Scale (MAAS) | at the entry into the study, and after 6 weeks
  a 15 item measure of mindfulness. The item content was design to reflect the opposite of the construct of mindfulness, or: "mindlessness" and thus endorsing the item content at a lower frequency is taken to represent a higher level of mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Pesach Shvartzman, M.D, Principal Investigator — Clalit Health Service
Locations (1):
- Clalit Health Service, Beersheba, Israel